CLINICAL TRIAL: NCT04163224
Title: Minimal Invasive Approach for Surgical Repair of Rib Fractures With a Novel Intrathoracic Device. Case Series
Brief Title: Minimal Invasive Approach for Surgical Repair of Rib Fractures With a Novel Intrathoracic Device
Acronym: RF-Advantage
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor strategy change
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 0719-2
Record Dates: First submitted 2019-11-08; First posted 2019-11-14 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Rib Fracture Multiple
Keywords: multiple rib fractures; chest stabilization; rib plates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: RibFix Advantage — Class II device in the United States; consists of bridges (with locking posts) and locking caps for the thoracoscopic fixation and stabilization of ribs. These implants are manufactured from commercially pure titanium and titanium alloys. When fully assembled, the bridge plate is placed on the underside of the rib (pleural cortex); the threaded locking posts extend through pre-drilled holes in the rib, and the locking caps are fixed to the locking post on the anterior (cutaneous) side of the rib. The combined threaded locking post and cap provides for fixation of the bridge and stabilization of the fracture.

SUMMARY:
A retrospective review of demographics and adverse events from cases completed with the RibFix Advantage System. Evaluation of device integrity, and performance by a prospective CT scan with a minimum of 3 months post-implantation.

DETAILED DESCRIPTION:
The RibFix Advantage System is a novel intrathoracic titanium plating system that is FDA-cleared for the treatment of rib fractures. The RibFix Advantage System is designed to be implanted in a less invasive procedure where plates are introduced and placed on the pleural cortex of the rib during video-assisted thoracoscopic surgery. Intrathoracic plate placement allows for smaller cutaneous incisions and less muscle disruption, which may aid in patient recovery compared to traditional open reduction internal fixation systems that are currently available.

The purpose of this study is to gather the first clinical data on this novel device in the context of a case series of patients with radiologic and quality-of-life follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* ≥ 18 years old (no upper limit)
* Underwent surgical repair of rib fracture(s) with the RibFix Advantage System alone or in combination with other systems for fracture repair
* Signed Informed Consent Form for participation in a clinical trial
* Willing and able to return for a follow-up visit (includes a computed tomography (CT) scan of the chest)

Exclusion Criteria:

* Off label use of RibFix Advantage (e.g., active or latent infection at the time of implantation, sepsis, metal sensitivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for rib fracture repair using RibFix Advantage System alone or in combination with other methods for rib fracture repair
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Fracture stability | 3 months post-implantation
  Evaluated by a computed tomography (CT) scan. Rib fractures repaired with RibFix Advantage should demonstrate continuity without overlap
Device integrity | 3 months post-implantation
  Evaluated by a computed tomography (CT) scan. Images should demonstrate no plate migration, no post/cap migration and no plate fracture

SECONDARY OUTCOMES:
Adverse Events of Interest | From the the date of implantation until the day of hospital discharge, or up to 10 days post-implantation, whichever occurs first; 30 days post surgery; 3 month post-implantation
  Includes: Chest infections, Empyema, Mediastinitis. Wound infection, Wound dehiscence, Chest wall deformity related to the device, Pleural effusion related to the device, Hemothorax related to the device, Pneumothorax related to the device and Hemo-pneumothorax related to the device

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sun, Study Director — Zimmer Biomet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Granetzny A, Abd El-Aal M, Emam E, Shalaby A, Boseila A. Surgical versus conservative treatment of flail chest. Evaluation of the pulmonary status. Interact Cardiovasc Thorac Surg. 2005 Dec;4(6):583-7. doi: 10.1510/icvts.2005.111807. Epub 2005 Sep 15. PMID 17670487
- [Background] Majercik S, Wilson E, Gardner S, Granger S, VanBoerum DH, White TW. In-hospital outcomes and costs of surgical stabilization versus nonoperative management of severe rib fractures. J Trauma Acute Care Surg. 2015 Oct;79(4):533-8; discussion 538-9. doi: 10.1097/TA.0000000000000820. PMID 26402525
- [Background] Pieracci FM, Agarwal S, Doben A, Shiroff A, Lottenberg L, Whitbeck SA, White TW. Indications for surgical stabilization of rib fractures in patients without flail chest: surveyed opinions of members of the Chest Wall Injury Society. Int Orthop. 2018 Feb;42(2):401-408. doi: 10.1007/s00264-017-3612-1. Epub 2017 Aug 29. PMID 28852836
- [Background] Sarani B, Allen R, Pieracci FM, Doben AR, Eriksson E, Bauman ZM, Gupta P, Semon G, Greiffenstein P, Chapman AJ, Kim BD, Lottenberg L, Gardner S, Marasco S, White T. Characteristics of hardware failure in patients undergoing surgical stabilization of rib fractures: A Chest Wall Injury Society multicenter study. J Trauma Acute Care Surg. 2019 Dec;87(6):1277-1281. doi: 10.1097/TA.0000000000002373. PMID 31107433
- [Result] Edwards JG, Clarke P, Pieracci FM, Bemelman M, Black EA, Doben A, Gasparri M, Gross R, Jun W, Long WB, Lottenberg L, Majercik S, Marasco S, Mayberry J, Sarani B, Schulz-Drost S, Van Boerum D, Whitbeck S, White T; Chest Wall Injury Society collaborators. Taxonomy of multiple rib fractures: Results of the chest wall injury society international consensus survey. J Trauma Acute Care Surg. 2020 Feb;88(2):e40-e45. doi: 10.1097/TA.0000000000002282. No abstract available. PMID 31590175
- [Result] Leinicke JA, Elmore L, Freeman BD, Colditz GA. Operative management of rib fractures in the setting of flail chest: a systematic review and meta-analysis. Ann Surg. 2013 Dec;258(6):914-21. doi: 10.1097/SLA.0b013e3182895bb0. PMID 23511840
- [Result] Majercik S, Cannon Q, Granger SR, Van Boerum DH, White TW. Regarding: Long-term patient outcomes after surgical stabilization of rib fractures. Am J Surg. 2015 Jul;210(1):199-200. doi: 10.1016/j.amjsurg.2015.03.020. Epub 2015 May 21. No abstract available. PMID 26072282
- [Result] Majercik S, Cannon Q, Granger SR, VanBoerum DH, White TW. Long-term patient outcomes after surgical stabilization of rib fractures. Am J Surg. 2014 Jul;208(1):88-92. doi: 10.1016/j.amjsurg.2013.08.051. Epub 2014 Jan 4. PMID 24507379
- [Result] Majercik S, Vijayakumar S, Olsen G, Wilson E, Gardner S, Granger SR, Van Boerum DH, White TW. Surgical stabilization of severe rib fractures decreases incidence of retained hemothorax and empyema. Am J Surg. 2015 Dec;210(6):1112-6; discussion 1116-7. doi: 10.1016/j.amjsurg.2015.08.008. Epub 2015 Sep 18. PMID 26454653
- [Result] Marasco SF, Davies AR, Cooper J, Varma D, Bennett V, Nevill R, Lee G, Bailey M, Fitzgerald M. Prospective randomized controlled trial of operative rib fixation in traumatic flail chest. J Am Coll Surg. 2013 May;216(5):924-32. doi: 10.1016/j.jamcollsurg.2012.12.024. Epub 2013 Feb 13. PMID 23415550
- [Result] Pieracci FM. Completely thoracoscopic surgical stabilization of rib fractures: can it be done and is it worth it? J Thorac Dis. 2019 May;11(Suppl 8):S1061-S1069. doi: 10.21037/jtd.2019.01.70. PMID 31205763
- [Result] Pieracci FM, Lin Y, Rodil M, Synder M, Herbert B, Tran DK, Stoval RT, Johnson JL, Biffl WL, Barnett CC, Cothren-Burlew C, Fox C, Jurkovich GJ, Moore EE. A prospective, controlled clinical evaluation of surgical stabilization of severe rib fractures. J Trauma Acute Care Surg. 2016 Feb;80(2):187-94. doi: 10.1097/TA.0000000000000925. PMID 26595710
- [Result] Pieracci FM, Majercik S, Ali-Osman F, Ang D, Doben A, Edwards JG, French B, Gasparri M, Marasco S, Minshall C, Sarani B, Tisol W, VanBoerum DH, White TW. Consensus statement: Surgical stabilization of rib fractures rib fracture colloquium clinical practice guidelines. Injury. 2017 Feb;48(2):307-321. doi: 10.1016/j.injury.2016.11.026. Epub 2016 Nov 27. No abstract available. PMID 27912931
- [Result] Slobogean GP, MacPherson CA, Sun T, Pelletier ME, Hameed SM. Surgical fixation vs nonoperative management of flail chest: a meta-analysis. J Am Coll Surg. 2013 Feb;216(2):302-11.e1. doi: 10.1016/j.jamcollsurg.2012.10.010. Epub 2012 Dec 5. PMID 23219148
- [Result] Tanaka H, Yukioka T, Yamaguti Y, Shimizu S, Goto H, Matsuda H, Shimazaki S. Surgical stabilization of internal pneumatic stabilization? A prospective randomized study of management of severe flail chest patients. J Trauma. 2002 Apr;52(4):727-32; discussion 732. doi: 10.1097/00005373-200204000-00020. PMID 11956391